CLINICAL TRIAL: NCT05812651
Title: Effects of Induced Inspiratory Muscle Fatigue on Functional Mobility of Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: REC/01375 Qurat ul ain Gohar
Record Dates: First submitted 2023-03-31; First posted 2023-04-13 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Healthy Older Adults
Keywords: Inspiratory muscle fatigue; Functional mobility; Maximum Inspiratory Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IMF arm (Experimental): The interventional protocol will include healthy older adults age above 60 years. At baseline - all measurements will be collected. After 3 days to one week, as per feasibility, participants will come to the lab again and perform inspiratory Muscle training according to the protocol that tends to induce inspiratory muscle fatigue. (60-80%MIP).
  Inspiratory resistive loading by starting at 60-80% (MIP) increasing every 10 minutes by 10% then measure Maximum Inspiratory Pressure (MIP), until MIP measurement decrease of more than 10% from baseline will be performed. When report a lower score of MIP and participants could no longer worked out, performed the functional mobility tests and see if there any variation. After the consent of participants an initial evaluation, Anthropometric measurements, Pulmonary function tests, PASE Questionnaire will be taken.
  Interventions: Other: Inspiratory muscle fatigue

INTERVENTIONS:
Other: Inspiratory muscle fatigue — Muscle training according to the protocol that tends to induce inspiratory muscle fatigue. (60-80% MIP). Inspiratory resistive loading by starting at 60-80% (MIP) increasing every 10 minutes by 10% then measure MIP, until MIP measurement decrease of more than 10% from baseline will be performed.
  When report a lower score of MIP and participants could no longer worked out, performed the functional mobility tests and see if there any variation.

SUMMARY:
The aim of study was to evaluate the effects of inspiratory induced muscle fatigue on functional mobility of older adults. Though, limited literature exists regarding inspiratory muscle fatigue and its consequences on functional activities of daily living and balance. Yet, it is not clear how improvement in inspiratory muscle strength is related with improvement in functional mobility.

DETAILED DESCRIPTION:
Respiratory muscle fatigue was first described in 1977. Inspiratory muscle relaxation rates are known to slow following induction of fatigue. Inspiratory muscle fatigue was induced by threshold loading at 80 percent of (Maximum Inspiratory Pressure) Pimax until the subjects were unable to generate the target pressure. Inspiratory muscle fatigue (IMF) is proposed to negotiation exercise performance, probably via a respiratory muscle metaboreflex that impairs blood flow to working muscles, thereby accelerating the progress of fatigue in these muscles. Respiratory muscle fatigue revealed that a maximal inspiratory load of 50% could quickly fatigue both the inspiration and expiration muscles. Increased inspiratory muscle work may induce fatigue of the respiratory muscles, as well as of the non-respiratory muscles by central alterations at spinal and supraspinal level. Also there is an association between respiratory muscle dysfunction and physical performance in older adults. The abnormalities of respiratory movements may be dependable clinical signs of inspiratory muscle fatigue, mostly when accompanied by tachypnea and hypercapnia. Fatigue is distinguished from weakness, a decrease in force generation that is static and not reversible by rest, though muscle weakness may be a susceptibility to muscle fatigue. This study will contribute to determine the effects of respiratory muscle fatigue on balance and functional mobility with healthy older adults. To further understand this relationship, a battery of tests (considered as gold standard) will be performed after induced inspiratory muscles fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Adults with age 60+ years
* Both male and female participants
* Patients with Forced Expiratory Volume 1/Forced Volume Capacity ratio greater than 80%

Exclusion Criteria:

* Smokers
* Subjects with a history of cardiovascular, respiratory, or neuromuscular
* Diseases that can impede test or alter the maximum inspiratory pressure.
* Subjects with cognitive impairment.
* Subjects with low back and musculoskeletal disorders.
* Previous experience in respiratory muscle training.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Six minute walk test | After 3 days
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance.
30sec sit to stand test | After 3 days
  The 30 Second Sit to Stand Test is also known as 30 second chair stand test ( 30CST), is for testing leg strength and endurance in older adults.
Arm curl field test | After 3 days
  The Arm Curl Fitness Test for upper body strength using the bicep curl technique, a test designed of the functional fitness of seniors
Stair climbing test | After 3 days
  The stair climb test (also known as stair climb power test) is a clinically relevant, safe, and inexpensive field-based assessment of lower body strength, power, and physical function for older adults

SECONDARY OUTCOMES:
Physical activity scale for elderly (PASE) | After 3 days
  Physical Activity Scale for the Elderly (PASE) is a brief (5 minutes) and easily scored survey designed specifically to assess physical activity in epidemiological studies of persons age 65 years and older. The PASE assesses the types of activities typically chosen by older adults (walking, recreational activities, exercise, housework, yard work, and caring for others. It uses frequency, duration, and intensity level of activity over the previous week to assign a score, ranging from 0 to 793, with higher scores indicating greater physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Suman Sheraz, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Railway General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seixas MB, Almeida LB, Trevizan PF, Martinez DG, Laterza MC, Vanderlei LCM, Silva LP. Effects of Inspiratory Muscle Training in Older Adults. Respir Care. 2020 Apr;65(4):535-544. doi: 10.4187/respcare.06945. Epub 2019 Oct 29. PMID 31662444
- [Background] Giua R, Pedone C, Scarlata S, Carrozzo I, Rossi FF, Valiani V, Incalzi RA. Relationship between respiratory muscle strength and physical performance in elderly hospitalized patients. Rejuvenation Res. 2014 Aug;17(4):366-71. doi: 10.1089/rej.2014.1549. PMID 24749768
- [Background] Watsford ML, Murphy AJ, Pine MJ. The effects of ageing on respiratory muscle function and performance in older adults. J Sci Med Sport. 2007 Feb;10(1):36-44. doi: 10.1016/j.jsams.2006.05.002. Epub 2006 Jun 30. PMID 16814604
- [Background] Ferraro FV, Gavin JP, Wainwright T, McConnell A. The effects of 8 weeks of inspiratory muscle training on the balance of healthy older adults: a randomized, double-blind, placebo-controlled study. Physiol Rep. 2019 May;7(9):e14076. doi: 10.14814/phy2.14076. PMID 31074198